CLINICAL TRIAL: NCT02974127
Title: Multisession Radiosurgery in Large Meningiomas
Acronym: MuRaLM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: SRS_LM
Record Dates: First submitted 2016-10-07; First posted 2016-11-28 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Intracranial Meningioma
Keywords: intracranial benign meningioma; radiosurgery; large meningioma; critical site; multisession radiosurgery
MeSH Terms: conditions — Meningioma | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy — Multisession radiosurgery
  Other Names: Radiosurgery

SUMMARY:
This is a prospective observational trial consisting of robotic multisession radiosurgery (CyberKnife ®) for large and medium size and/or located at critical site benign intracranial meningiomas.

DETAILED DESCRIPTION:
To date, the treatment of choice for intracranial meningiomas is surgical removal.

Radiotherapy, especially the radiosurgery (SRS), in exclusive, adjuvant or salvage setting represents an alternative or complementary viable treatment to the neurosurgery. Despite being a well-established treatment for intracranial meningiomas, SRS might be associated with significant morbidity when large volumes or critical sites are treated. Hypofractionated stereotactic radiotherapy has the potential to deliver sharply focused high doses per fraction without increasing the risk of toxicity.

The aims of our study are toxicity and symptom control evaluation of radiosurgery treatment delivered in multisession, for large or medium size intracranial meningiomas and/or for intracranial meningioma located at the critical sites (perichiasmatic area, perioptic area, PCA). We will evaluate also the efficacy of the treatment by volumetric analysis of treated meningiomas carrying out a volumetric comparison between pre- and post-radiosurgery treatment (every 6 month after treatment).

The neurological and clinical assessment before and after s-SRS will be based on CTCAE v4.0 and BPN BSN House-Brackman and sensorineural internation scale assessment.

ELIGIBILITY:
Inclusion Criteria:

* either histologically confirmed or imaging-defined benign meningioma diagnosis;
* large or medium lesion size and/or in critical area (e.i. perichiasmatic area);
* signed specific informed consent;
* age ≥ 18 years;
* for female patients, execution of pregnancy blood test;
* Karnofsky Performance Status (KPS) ≥ 70.

Exclusion Criteria:

* histologically confirmed diagnosis of atypical or malignant meningiomas;
* patients who had received prior radiotherapy in the same site;
* pregnancy;
* allergy for contrast medium;
* neurofibromatosis diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large or in critical site benign intracranial meningioma diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Radiation-related toxicities. | change from baseline neurological assessment at 5 years.
  evaluation every 6 months, up to 3 years. Afterwards, every year up to 5 years based on CTCAE v4.0
Local control evaluation assessed on MRI-based volumetric lesion measurements. | change from baseline volume lesion at 5 years
  Evaluation based on 1-3 mm thickness T1 weighted (or volumetric FAT saturation weighted) brain gadolinium-MRI images

SECONDARY OUTCOMES:
Neurological assessment of trigeminal pain | every 6 months, up to 3 years. Afterwards, every year up to 5 years.
  Evaluation based on BNP scale
Neurological assessment of trigeminal dysfunction | every 6 months, up to 3 years. Afterwards, every year up to 5 years.
  Evaluation based on BNS scale
Neurological assessment of facial nerve dysfunction | every 6 months, up to 3 years. Afterwards, every year up to 5 years.
  Evaluation based on House-Brackman scale
Neurological assessment of acoustic nerve dysfunction | every 6 months, up to 3 years. Afterwards, every year up to 5 years.
  Evaluation based on sensorineural international scale
Neurological assessment of visual dysfunction | every 6 months, up to 3 years. Afterwards, every year up to 5 years.
  Evaluation based on ophthalmological evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fariselli, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo BEsta
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Unit of Radiotherapy, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pinzi V, Marchetti M, Viola A, Tramacere I, Cane I, Iezzoni C, Fariselli L. Hypofractionated Radiosurgery for Large or in Critical-Site Intracranial Meningioma: Results of a Phase 2 Prospective Study. Int J Radiat Oncol Biol Phys. 2023 Jan 1;115(1):153-163. doi: 10.1016/j.ijrobp.2022.08.064. Epub 2022 Sep 6. PMID 36075299
- [Derived] Pinzi V, Marchetti M, De Martin E, Cuccarini V, Tramacere I, Ghielmetti F, Fumagalli ML, Iezzoni C, Fariselli L. Multisession radiosurgery for intracranial meningioma treatment: study protocol of a single arm, monocenter, prospective trial. Radiat Oncol. 2020 Jan 30;15(1):26. doi: 10.1186/s13014-020-1478-7. PMID 32000819